CLINICAL TRIAL: NCT06898372
Title: Multicenter Retrospective Observational Study to Evaluate the Efficacy of Anti-Jak1 Inhibitors as Treatment for Patients With Aicardi-Goutières Syndrome
Brief Title: Evaluate the Efficacy of Anti-Jak1 Inhibitors as Treatment for Patients With Aicardi-Goutières Syndrome
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Roberta Battini, PHD, Professor, Medical Doctor, IRCCS Fondazione Stella Maris
Other Study IDs: AGS-AntiJak1
Record Dates: First submitted 2025-03-05; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Aicardi-Goutières Syndrome (AGS)
Keywords: Anti-Jak1/2; Ruxolitinib; Baricitinib; AGS-related interferonopathies
MeSH Terms: interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AAGS or AGS-related interferonopathies treated with Anti-Jak1/2: Study group:
  1. Patients aged 0 to 25 years
  2. Genetic diagnosis of Aicardi-Goutières Syndrome or AGS-related interferonopathies
  3. Treatment with Janus Kinase 1/2 (JAK1/2) inhibitors, including Baricitinib and Ruxolitinib
  Interventions: Drug: JAK Inhibitor
- Patients with AGS or AGS-related interferonopathies not treated with Anti-Jak1/2: Control group:
  1. Patients aged 0 to 25 years matched with the study cases
  2. Genetic diagnosis of Aicardi-Goutières Syndrome or AGS-related interferonopathies with genotype matched to the study cases
  3. Not treated with Janus Kinase 1/2 (JAK1/2) inhibitors, such as Baricitinib and Ruxolitinib

INTERVENTIONS:
Drug: JAK Inhibitor — The retrospective analysis will examine the effects of Janus Kinase 1/2 (JAK1/2) inhibitors, such as Baricitinib and Ruxolitinib, on neurological symptoms and brain MRI.
  Groups: Patients with AAGS or AGS-related interferonopathies treated with Anti-Jak1/2

SUMMARY:
Aicardi-Goutières Syndrome (AGS) is a hereditary multisystem autoinflammatory disorder that predominantly affects the central nervous system. It is characterized by severe neurological disability and chronic inflammation caused by the persistent overproduction of type I interferon. To date, nine causative genes of AGS have been identified, each of which can lead to classic AGS presentations, atypical forms, or other manifestations that do not meet the formal diagnostic criteria for AGS and are referred to as "AGS-related interferonopathies." Janus Kinase 1 (JAK1) inhibitors, including Baricitinib and Ruxolitinib, offer a promising therapeutic strategy for Aicardi-Goutières Syndrome (AGS) by directly targeting the central pathogenic pathway of the disease.

Patients treated with JAK1 inhibitors for AGS have shown significant improvement in systemic symptoms, though the effect on neurological symptoms and brain imaging remains unclear.

The aim of this project is to retrospectively analyze the efficacy, particularly on neurological symptoms and brain imaging, and the safety of JAK1 inhibitor treatment in AGS patients treated at Italian tertiary centers. Data will be collected before starting the therapy and during follow-up at 6, 12, 18, and 24 months, where available.

Preliminary data collection was carried out through a survey conducted by the AGS Italy group to assess the number of patients treated with JAK1 inhibitors.

Clinical, brain imaging, genetic, and laboratory data routinely recorded in nine different Italian centers as part of the standard clinical care of these patients will be retrospectively collected and analyzed.

In the second phase of the study, brain MRI data from AGS patients treated with JAK1 inhibitors will be compared to untreated AGS patients matched for age and genotype, in order to evaluate the potential therapeutic efficacy of JAK1 inhibitors on brain imaging compared to the natural clinical progression of the disease.

Through the analysis of the Italian experience, this study could lay the groundwork for drafting a potential consensus on the use of JAK1 inhibitors for the treatment of AGS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 25 years
* Patients who have been genetically diagnosed with Aicardi-Goutières Syndrome (AGS) or AGS-related interferonopathies For case cohort-Patients treated with Janus Kinase 1/2 (JAK1/2) inhibitors, such as Baricitinib or Ruxolitinib

Exclusion Criteria:

* Patients over the age of 25 years
* Patients who have not been genetically diagnosed with Aicardi-Goutières Syndrome (AGS) or AGS-related interferonopathies.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of approximately 24 patients with Aicardi-Goutières Syndrome or AGS-related interferonopathies are expected to be enrolled, including 12 patients treated with different Janus Kinase 1/2 (JAK1/2) inhibitors, such as Baricitinib and Ruxolitinib, and 12 untreated patients, from the 9 Italian clinical centers involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of JAK-1/2 inhibitor therapy on Clinical criteria (AGS scale) | After 6, 12, 18, and 24 months of treatment, if the data is available.
  Evaluate the efficacy of JAK-1/2 inhibitor therapy through clinical criteria (AGS scale) in all patients with Aicardi-Goutières Syndrome or AGS-related interferonopathies, highlighting potential differences in efficacy between the different genotypes. The Aicardi-Goutières Syndrome (AGS) Severity Scale is a clinical tool used to assess the severity of neurological impairment in individuals with AGS. The scale ranges from 0 to 11, with higher scores indicating better neurological function.
Efficacy of JAK-1/2 inhibitor therapy on laboratory parameter (IFN signature) | After 6, 12, 18, and 24 months of treatment, if the data is available.
  Evaluate the efficacy of JAK-1/2 inhibitor therapy through IFN signature (IFN score) on blood in all patients with Aicardi-Goutières Syndrome or AGS-related interferonopathies, highlighting potential differences in efficacy between the different genotypes. The IFN Score is typically expressed as a fold change relative to healthy controls or as a normalized relative value, measuring the expression of interferon-stimulated genes (ISGs). In patients with pathological activation of the interferon pathway, the IFN Score ranges from 0 to >10-15, indicating significant ISG upregulation. While the pathological cut-off varies across studies, an IFN Score >2-3 is often considered indicative of abnormal interferon pathway activation.
Efficacy of JAK-1/2 inhibitor therapy on instrumental parameters (brain MRI) | After 6, 12, 18, and 24 months of treatment, if the data is available.
  Evaluate the efficacy of JAK-1/2 inhibitor therapy through brain MRI (Improved/Unchanged/Worsening) in all patients with Aicardi-Goutières Syndrome or AGS-related interferonopathies, highlighting potential differences in efficacy between the different genotypes.
Evaluate the side effects of JAK-1/2 inhibitor | After 6, 12, 18, and 24 months of treatment, if the data is available.
  Evaluate the side effects of JAK-1/2 inhibitor therapy in patients with Aicardi-Goutières Syndrome or AGS-related interferonopathies.

SECONDARY OUTCOMES:
Consensus on indication of JAK-1/2 Inhibitor Therapy for Aicardi-Goutières Syndrome and Related Interferonopathies on Clinical criteria (AGS scale) | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on AGS scale criteria that define the indication for starting JAK-1/2 inhibitor therapy in Aicardi-Goutières Syndrome or AGS-related interferonopathies. The Aicardi-Goutières Syndrome (AGS) Severity Scale is a clinical tool used to assess the severity of neurological impairment in individuals with AGS. The scale ranges from 0 to 11, with higher scores indicating better neurological function.
Consensus on indication of JAK-1/2 Inhibitor Therapy for Aicardi-Goutières Syndrome and Related Interferonopathies on genetic criteria (type of Genetic mutation) | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on Genetic mutation that define the indication for starting JAK-1/2 inhibitor therapy in Aicardi-Goutières Syndrome or AGS-related interferonopathies. At now nine causative genes for Aicardi-Goutières Syndrome (AGS) are known: TREX1, RNASEH2A, RNASEH2B, RNASEH2C, SAMHD1, ADAR1, IFIH1, LSM11, and RNU7-1, all involved in nucleic acid metabolism and the interferon pathway.
Consensus on indication of JAK-1/2 Inhibitor Therapy for Aicardi-Goutières Syndrome and Related Interferonopathies on laboratory parameter (IFN signature) | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on laboratory parameter (IFN signature) that define the indication for starting JAK-1/2 inhibitor therapy in Aicardi-Goutières Syndrome or AGS-related interferonopathies.
  The IFN Score is typically expressed as a fold change relative to healthy controls or as a normalized relative value, measuring the expression of interferon-stimulated genes (ISGs). In patients with pathological activation of the interferon pathway, the IFN Score ranges from 0 to >10-15, indicating significant ISG upregulation. While the pathological cut-off varies across studies, an IFN Score >2-3 is often considered indicative of abnormal interferon pathway activation.
Consensus on Monitoring laboratory parameter (IFN signature) for JAK-1/2 Inhibitor Therapy in Aicardi-Goutières Syndrome and Related Interferonopathies | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on laboratory parameter (IFN signature) to be monitored during JAK-1/2 inhibitor therapy to assess the potential continuation or discontinuation due to lack of efficacy. The IFN Score is typically expressed as a fold change relative to healthy controls or as a normalized relative value, measuring the expression of interferon-stimulated genes (ISGs). In patients with pathological activation of the interferon pathway, the IFN Score ranges from 0 to >10-15, indicating significant ISG upregulation. While the pathological cut-off varies across studies, an IFN Score >2-3 is often considered indicative of abnormal interferon pathway activation.
Consensus on Monitoring Clinical criteria (AGS scale) for JAK-1/2 Inhibitor Therapy in Aicardi-Goutières Syndrome and Related Interferonopathies | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on Clinical criteria (AGS scale) to be monitored during JAK-1/2 inhibitor therapy to assess the potential continuation or discontinuation due to lack of efficacy. The Aicardi-Goutières Syndrome (AGS) Severity Scale is a clinical tool used to assess the severity of neurological impairment in individuals with AGS. The scale ranges from 0 to 11, with higher scores indicating better neurological function.
Consensus on instrumental parameters (brain MRI) for JAK-1/2 Inhibitor Therapy in Aicardi-Goutières Syndrome and Related Interferonopathies | Until study completion, an average of 2 year.
  Develop a possible consensus within the AGS Italia network on brain MRI to be monitored during JAK-1/2 inhibitor therapy to assess the potential continuation or discontinuation due to lack of efficacy. Evaluate based on the progression of brain MRI to determine whether it improves, remains stable, or worsens.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Stella Maris Foundation, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
A common format (Case Report Form, CRF) for all the centers involved in the study will be used to record data for each enrolled patient. In addition, all data related to the study have been and will be shared through a mailing list.
Supporting Information: Study Protocol, SAP, ICF, CSR